CLINICAL TRIAL: NCT00220675
Title: Recombinant Human Erythropoietin (r-HuEPO) in the Prevention of Neurologic Sequelae From Malignant Spinal Cord Compression: a Multi-Center, Placebo-Controlled, Phase 2 Randomized Study
Brief Title: Erythropoietin Spinal Cord Compression Randomized Trial
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Dr. Andrew Loblaw, Sunnybrook & Women's College Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9427-T0926-28C
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Nerve Compression Syndromes
Keywords: Malignant extradural spinal cord compression; Erythropoietin; Neuroprotectant; Radiotherapy; Palliation
MeSH Terms: conditions — Nerve Compression Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Erythropoietin infusion

SUMMARY:
To determine whether erythropoietin, steroids and radiotherapy is safe and feasible to administer to patients with malignant spinal cord compression.

DETAILED DESCRIPTION:
For patients with malignant spinal cord compression (MSCC) who are paraparetic or paraplegic before initiating treatment, the current treatment options provide a meager to poor chance of neurologic recovery and the prognosis is guarded. Improving the chance of ambulation after treatment for MSCC may dramatically improve patients' quality of life, decrease days spent in hospital and improve survival. Steroids appear to prevent neurologic damage from MSCC and increasing doses appear to have an increasingly protective effect, however, higher doses are limited by an increasing incidence of serious toxicity.

Recombinant human erythropoetin has been shown to improve quality of life in patients with anemia of chronic disease and animal models suggest that r-HuEPO may have a neuroprotective effect. Human studies have demonstrated increased CSF concentrations of r-HuEPO after intravenous administration, including patients with MESCC. Furthermore, there is a suggestion that patients treated with intravenous r-HuEPO, steroids and RT may recover ambulatory function to a greater degree and faster than patients not treated with r-HuEPO.

Ultimately the effect of r-HuEPO in improving neurologic, functional and quality of life outcomes will need to be tested in a properly designed, large, randomized control trial. However, in order to successfully complete this study in a timely manner, a multicenter study will need to be performed. There are logistical issues that need to be addressed when setting up a r-HuEPO infusion program.

Therefore, a multicenter, randomized phase 2 study of intravenous r-HuEPO, steroids and RT will allow the investigators to address three issues: i) confirm that the logistical issues at each center can be addressed; ii) confirm in a larger cohort of patients whether the encouraging neurologic outcomes seen in the preliminary study can be replicated across different settings when compared with a randomized control group; iii) ensure the safety of EPO in this population including overall survival and incidence of subsequent TVEs with and without EPO.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years old) with histopathologically confirmed cancer
* Patients unable to ambulate independently due to paraparesis or paraplegia from malignant epidural spinal cord compression (categories 2, 3, 4 in Appendix B)
* Radiotherapy offered for treatment of cord compression using 2000cGy in 5 fractions
* Informed consent signed
* Females subjects must be post-menopausal or surgically incapable of childbearing potential, must be practicing an acceptable method of birth control (i.e., hormonal contraceptives, intrauterine device or barrier and spermicide)

Exclusion Criteria:

* Uncontrolled hypertension (systolic pressure > 160 mmHg, diastolic > 100 mmHg) or unstable cardiovascular disease
* Previous DVT/PE or arterial embolic event
* Patients with a Hb > 120 g/L or Hct > 40% (for both males & females)
* Patients with potentially curable disease
* Patients with life expectancy < 3 months
* Patients who have received RT that would overlap with the planned treatment field
* Contraindications for MRI scan
* Women who are pregnant, or who intend to become pregnant, or who are nursing
* Patients with known brain metastases; those with a primary diagnosis of melanoma will require confirmation by CT or MRI
* Patients with a history of poorly controlled seizure disorder
* Patients with a known hypersensitivity to mammalian cell-derived products or albumin
* Patients who cannot receive adequate antithrombotic treatment, who have a hypersensitivity to the active antithrombotic substance or any of the product's excipients
* Patients who have participated in another investigational device or drug trial(s), or is receiving other investigational agent(s) within the previous 30 days
* Patients requiring neurosurgical decompression for the malignant spinal cord compression

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Overall survival
Recovery of ambulation
Deep vein thrombosis rate post-treatment

SECONDARY OUTCOMES:
The time to regain ambulation
Duration of ambulatory function
Health-related quality of life (HRQOL, prevalence of TVE at the time of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, MD MSc, Principal Investigator — Sunnybrook & Women's College Health Science Centre
Locations (3):
- Canada (3):
  - London Regional Health Science Center, London, Ontario
  - Ottawa Regional Cancer Center, Ottawa, Ontario
  - Sunnybrook & Women's College Health Science Centre, Toronto, Ontario